CLINICAL TRIAL: NCT06453538
Title: Sleep Quality and Sleep-disordered Breathing in Bypass Surgery Patients
Acronym: UNI-CABG
Status: Recruiting | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Marjo Ajosenpää, Principal Investigator, Turku University Hospital
Other Study IDs: 27 /1801/2022
Record Dates: First submitted 2024-04-10; First posted 2024-06-11 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Sleep Disorder; Coronary Artery Disease
MeSH Terms: conditions — Sleep Wake Disorders; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients undergoing non-emergency coronary artery bypass surgery (CABG) are included. All patients will be examined for transthoracic echo, blood samples will be collected, and an overnight sleep polygraph will be performed in a qualified sleep laboratory twice: once before CABG and again after surgery

DETAILED DESCRIPTION:
Detailed Description:

Our hypothesis is that sleep-related apneas are increasing following coronary artery bypass surgery, and sleep quality may deteriorate. We are attempting to determine the causes of these difficulties, which are caused by microemboli in the brain from the use of a heart-lung machine, brain infarction induced by major surgery, thoracic tissue trauma following surgery, or complications during perioperative care. The hypothesis is that postoperative outcomes and recovery are related if a patient is identified with sleep apnea before CABG surgery. A sleep polygraph is performed before surgery and again around six months after, as well as a transthoracic echo and laboratory tests. If a link between sleep quality and coronary bypass surgery can be established, the results can be employed in clinical practice.

The total amount of patients operated on heart-lung machine is anticipated to be 70. The off-pump patient sample size is remarkably smaller, so data is collected and compared with the main sample population. The operation technique is decided when the patient is scheduled for operation. Emergency patients are excluded because pre-operative examinations cannot be performed. Other exclusion criteria are nighttime CPAP- treatment and other heart operations (for example valve surgery) during CABG.

Basic information including age, weight, height, diseases, medications, and medical history are collected from all patients. ECG is registered before and after surgery and sinus or other heart rhythms are recorded. Sleep polygraph is done preoperatively and postoperatively when the patient is fully recovered from surgery (at 6 months or more).

ELIGIBILITY:
Inclusion Criteria:

Elective coronary artery bypass surgery

Exclusion Criteria:

* Emergency cabg
* Night time cpap- treatment
* other heart operations (for example valve surgery)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All scheduled volunteered coronary artery bypass patients in Turku University Hospital area
Sampling Method: Non-Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of sleep disorders before coronary artery bypass surgery (CABG), polysomnography | Before operation, as soon as operation has scheduled
  Apnea-hypopnea index (AHI). Number of apneas and hypopneas that occur per hour of sleep. According to the American Academy of Sleep Medicine (AASM) it is categorized into mild (5-15 events/hour), moderate (15-30 events/hr), and severe (> 30 events/hr) (1).
Sleep quality before CABG | Before operation, as soon as operation has scheduled
  ESS, EPWORTH SLEEPINESS SCALE. All scores on the Epworth Sleepiness Scale fall between 0 and 24. Scores from 0 to 10 reflect normal levels of daytime sleepiness, and scores over 10 are considered to reflect excessive daytime sleepiness.
A transthoracic echocardiogram | Before operation, as soon as operation has scheduled
  Left ventricular end-diastolic diameter (LVEDD), Left ventricular end-systolic diameter (LVESD), Septal wall thickness (SWT), and Posterior wall thickness (PWT), Max/Min Diameter of IVC; all will be reported in cm.

SECONDARY OUTCOMES:
Incidence of sleep disorders after coronary artery bypass surgery, polysomnography | After 6 to 8 months after surgery
  Apnea-hypopnea index (AHI). Number of apneas and hypopneas that occur per hour of sleep. According to the American Academy of Sleep Medicine (AASM) it is categorized into mild (5-15 events/hour), moderate (15-30 events/hr), and severe (> 30 events/hr) (1).
Sleep quality after CABG | After 6 to 8 months after surgery
  ESS, EPWORTH SLEEPINESS SCALE. All scores on the Epworth Sleepiness Scale fall between 0 and 24. Scores from 0 to 10 reflect normal levels of daytime sleepiness, and scores over 10 are considered to reflect excessive daytime sleepiness
A transthoracic echocardiogram | After operation, 3-5 months after surgery
  Left ventricular end-diastolic diameter (LVEDD), Left ventricular end-systolic diameter (LVESD), Septal wall thickness (SWT), and Posterior wall thickness (PWT), Max/Min Diameter of IVC; all will be reported in cm.

OTHER OUTCOMES:
New York Heart Association -classification (NYHA) status | Before operation
  Class I - No symptoms and no limitation in ordinary physical activity, e.g. shortness of breath when walking, climbing stairs etc.
  Class II - Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity.
  Class III - Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20-100 m).Comfortable only at rest.
  Class IV - Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients

CONTACTS AND LOCATIONS:
Overall Officials: Nea Kalleinen, millä Associate Professor, Study Director — Turku University Hospital/Heart Center
Locations (1):
- Turku University Hospital, Turku, Finland

IPD SHARING:
Plan to Share IPD: No